CLINICAL TRIAL: NCT04143555
Title: Prospective Registry Study of Endoscopic Submucosal Injection of Indocyanine Green Before Laparoscopic Gastrectomy
Brief Title: Endoscopic Submucosal Injection of Indocyanine Green Before Laparoscopic Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Dong Yang, Doctor, Jilin University
Other Study IDs: 130002
Record Dates: First submitted 2019-10-27; First posted 2019-10-29 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Endoscopic Submucosal Injection of Indocyanine Green
Keywords: endoscopic submucosal injection; indocyanine green

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endoscopic submucosal injection of indocyanine green
  Interventions: Procedure: endoscopic submucosal injection of indocyanine green before laparoscopic gastrectomy

INTERVENTIONS:
Procedure: endoscopic submucosal injection of indocyanine green before laparoscopic gastrectomy — Indocyanine green was injected under endoscope within 24 hours before operation. Four points(0.5ml/point,1.25mg/ml) were evenly injected in four quadrants at the edge of the tumor. The injection method was direct submucosal injection and 0.5ml saline + 0.5ml indocyanine green solution + 0.5ml saline (sandwich method). The imaging effect was evaluated by indocyanine green fluorescence imaging system during the operation. The effect was divided into grade0 and Grade1. Grade1: The imaging of the tumor and the corresponding lymphatic drainage area in the injection area both were ideal. Grade 0: not up to grade 1, classified into tumor body and drainage area without imaging, only tumor body imaging, and even though tumor body and regional lymph drainage area imaging, the contrast agent in the gastric wall was too diffuse or even overflowing, which seriously interfered with the observation of lymph drainage area imaging.

SUMMARY:
Prospective registry study of endoscopic submucosal injection of indocyanine green before laparoscopic gastrectomy

DETAILED DESCRIPTION:
To observe the imaging result of endoscopic submucosal injection of indocyanine green before laparoscopic gastrectomy, and analyze the relevant factors, so as to guide the operation of preoperative indocyanine green submucosal injection better.

This study is prospective and observational. In order to analyze the related factors that affect the imaging effect, we enrolled patients who were to undergo indocyanine green fluorescence imaging for laparoscopic radical gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients who were to undergo indocyanine green fluorescence imaging for laparoscopic radical gastrectomy.

Exclusion Criteria:

* have simultaneously other cancer

  * have severe systemic inflammatory disease ,serious illness such as diabetes, chronic lung diseases
  * have upper gastrointestinal surgery
  * Indocyanine green or iodine allergy
  * the period is too late or the tumor is too large to carry on a laparoscopy assisted radical distal gastrectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were to undergo indocyanine green fluorescence imaging for laparoscopic radical gastrectomy for gastric cancer
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-04-10 (Estimated); Study Completion 2021-04-20 (Estimated)

PRIMARY OUTCOMES:
The imaging effect of indocyanine green | During the operation
  The imaging effect was evaluated by indocyanine green fluorescence imaging system during the operation. The effect was divided into grade0 and Grade1. Grade1: The imaging of the tumor and the corresponding lymphatic drainage area in the injection area both were ideal. Grade 0: not up to grade 1, classified into tumor body and drainage area without imaging, only tumor body imaging, and even though tumor body and regional lymph drainage area imaging, the contrast agent in the gastric wall was too diffuse or even overflowing, which seriously interfered with the observation of lymph drainage area imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No